CLINICAL TRIAL: NCT01688518
Title: Evaluation of the Depth and Duration of Anesthesia From Heated Lidocaine/Tetracaine (Synera®) Patches Compared With 5% Lidocaine (Lidoderm®) Patches Applied to Healthy Adult Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: CRI Lifetree (Other)
Collaborators: Nuvo Research Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: LCR-07-01-101
Record Dates: First submitted 2012-09-17; First posted 2012-09-20 (Estimated); Last update posted 2013-01-04 (Estimated); Status verified 2013-01

CONDITIONS: Healthy
Keywords: Evaluation; Depth and Duration; Anesthesia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Synera® for 30min & Lidoderm® for 4 hours (Active Comparator): Heated Lidocaine/Tetracaine (Synera®)applied to one forearm for either 30 minutes or 4 hours and a 5% Lidocaine (Lidoderm®) patch applied to the alternate forearm for the alternate time period.
  Interventions: Drug: Heated Lidocaine/Tetracaine Patch; Drug: 5% Lidocaine Patch
- Lidoderm® for 30min & Synera® for 4 hours (Active Comparator): Heated Lidocaine/Tetracaine (Synera®)applied to one forearm for either 30 minutes or 4 hours and a 5% Lidocaine (Lidoderm®) patch applied to the alternate forearm for the alternate time period.
  Interventions: Drug: Heated Lidocaine/Tetracaine Patch; Drug: 5% Lidocaine Patch

INTERVENTIONS:
Drug: Heated Lidocaine/Tetracaine Patch
  Other Names: Synera® Patch
Drug: 5% Lidocaine Patch
  Other Names: Lidoderm® Patch

SUMMARY:
This will be a randomized, single-blind, active-controlled, two-period crossover study in adult volunteers to compare the duration and depth of anesthesia between Synera® and Lidoderm® patches when applied for 30 minutes and 4 hours. The study will include a Screening Visit, two Treatment Periods, and a Follow-Up Phone Contact.

ELIGIBILITY:
Inclusion:

1. Subject is male or female 18-60 years of age, inclusive.
2. Subject is judged by the Investigator to be in generally good health at screening based upon the results of a medical history, physical examination, clinical laboratory profile, and 12-lead electrocardiogram (ECG).
3. Subject is willing to refrain from using any local topical preparations on the volar aspect of the forearms for 24 hours prior to each site visit.
4. Subject has normal, intact skin bilaterally at the antecubital area.
5. If female, must be of non-childbearing potential (defined as postmenopausal for at least 1 year or surgically sterile [bilateral tubal ligation, bilateral oophorectomy or hysterectomy]) or must be using adequate contraception (practicing one of the following methods of birth control):

   * Total abstinence from sexual intercourse (minimum of one complete menstrual cycle before study entry),
   * A vasectomized partner,
   * Contraceptives (oral, parenteral, or transdermal) for 3 consecutive months prior to test product administration,
   * Intrauterine device (IUD), or
   * Double-barrier method (condoms, sponge, diaphragm, or vaginal ring with spermicidal jellies or cream).
6. If female, must have a negative urine pregnancy test at Screening and at check-in of each Treatment Period.
7. Subject is willing to be blindfolded during the study and agrees to abide by all study restrictions and comply with all study procedures.
8. Able to fluently speak and understand English and be able to provide meaningful written informed consent for the study.

Exclusion:

1. Subject has clinically significant ECG abnormalities at screening.
2. Subject is currently receiving class I, II, or III anti-arrhythmic agents.
3. Subject has used over-the-counter (OTC) or prescription analgesics within 24 hours prior to either study period.
4. Subject has a known allergy or history of significant adverse reaction to any component of the treatment or related compounds.
5. Subject has a history of or active use or abuse of illicit drug substance or alcohol abuse.
6. Subject has a positive urine test result for drugs of abuse or a positive ethanol breath test at the Screening Visit or check-in to Treatment Visit 1.
7. Subject has active dermatological disease of any origin that may interfere with the ability to participate.
8. Subject has denuded or broken skin on either forearm.
9. Subject has a history of unstable peripheral/vascular disease and/or hypertensive vascular disease.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2012-09; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Depth of Anesthesia measured in mm via insertion of 21-gauge needle into the skin. | Approximately 5 months

SECONDARY OUTCOMES:
Duration of Anesthesia measured in sensory presence, absence, and thermal thresholds. | Approximately 5 months

CONTACTS AND LOCATIONS:
Overall Officials: Miroslav Backonja, MD, Principal Investigator — CRI Lifetree
Locations (1):
- Lifetree Clinical Research, Salt Lake City, Utah, United States